CLINICAL TRIAL: NCT04414436
Title: A Guided Internet Intervention for Women Treated for Gynecological Cancer
Acronym: GYNEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); VID Specialized University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9612
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Quality of Life
Keywords: cancer
MeSH Terms: conditions — Neoplasms | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: active intervention group vs waiting list group. Waitling list group crossing over to active group after 6 weeks
Who Masked: Participant
Masking Description: study participants will be identified with an anonymous ID
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GYNEA- digital coping program (Experimental): Participants randomized to this arm will receive active treatment after the inclusion
  Interventions: Behavioral: GYNEA- digital coping program for women after gynaecological cancer
- Waiting list (No Intervention): 6 weeks waiting list before crossing over to GYNEA- digital coping program

INTERVENTIONS:
Behavioral: GYNEA- digital coping program for women after gynaecological cancer — 6 modules with relevant information and tools for coping after cancer
  Other Names: waiting list
  Arms: GYNEA- digital coping program

SUMMARY:
Gynecological cancers are the sixth most common cancer forms and the number of survivors is increasing as a consequence of more efficient treatment and longer life span. As part of regulary care after cancer treatment the women have five years of follow-up with the primary focus on recurrence, aiming to increase survival. However, several studies have shown that there is no evidence for this assumption on increased survival (ref). There are now suggested alternative perspectives in the follow up period targeting late effects, health-related quality of life (QoL) and patient satisfaction with care.The main aim of the current study is to test the feasibility and acceptability of an internet-based psychosocial intervention for women treated with curative intent gynecological cancer. Another aim is to test the perceived effect on gynecological cancer survivors health-related self-care and QoL.

DETAILED DESCRIPTION:
The study's objectives and research questions Research questions

1. How did the participants use the program?

   1. What are the barriers and facilitators concerning technologies of the internet-based self -management intervention?
   2. Number of logins
   3. How much time did the participants spend on the program (per login )
   4. Number of modules completed, number of home-work and mindfulness assignment completed
   5. Type of errors made …
2. What is the participants' perceived credibility of the program?
3. How do the participants experience the guided psychosocial digital intervention?

   1. How do participants experience the cancer trajectory, their every-day lives and health-related QoL post-treatment gynaecological cancer (before the intervention)?
   2. How do the participants experience the internet-based intervention regarding content, the home-work assignments, and the mindfulness assignments, the active participation?
   3. How do the participants experience the telephone-contact and follow-ups with the nurse once a week?
   4. Which factors do they describe as important for their satisfaction and dissatisfaction
4. How is the perceived effect on the gynecological cancer survivors' competence, QoL, self-care and coping?

It is hypothesized that an internet-based psycho-social intervention will support women in developing self-competence and self-care which could be measured as increased QOL and secondarily affect the impact of cancer, distress, anxiety, depression, self-esteem, and self-reported ability to monitor and respond to symptoms of recurrence.

ELIGIBILITY:
Inclusion Criteria

* have had gyneocological cancer
* maximum 1 year after gynecological cancer

Exclusion Criteria:

* severe medical or psychiatric condition
* relapse of gynecological cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gyneocological cancer
Enrollment: 100 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The Impact of Cancer version 2 | up to 26 weeks
  Designed to assess the physical and psychosocial health experience of cancer survivors through its positive and negative impacts. 47-item questionnaire organized into 4 positive (altruism and empathy (AE), health awareness (HA), meaning of cancer (MOC), positive self-evaluation (PSE)) and 4 negative (appearance concerns (AC), body change concerns (BCC), life interference (LI) and worry (W)) impact dimensions [13] corresponding to the first 37 items. The questionnaire also includes 10 additional items constituting conditional dimensions applicable to subsets of survivors assessing employment concerns (EC), relationship concerns for individuals with a partner (P), and relationship concerns for those without a partner (NP). All items are scored on a five-point scale from 1 = strongly disagree to 5 = strongly agree. A higher score on a dimension implies stronger endorsement of that content area
The Quality of Life Patient/Cancer Survivor Version | up to 26 weeks
  ordinal questionnaire measuring the quality of life in cancer patients over 42 items rated on 10 point Likert-type scale. The revised instrument included 41 items representing the four domains of quality of life incorporating physical, psychological, social, and spiritual well being.
Patient Health Questionnaire | up to 26 weeks
  Subjects indicated for each of the nine depressive symptoms (corresponding to the criteria ofDSM-IV) whether, during the previous 2 weeks, the symptom has bothered them: 0=not at all; 1=several days; 2=more than half of the days; 3=nearly every day.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Bergen Municipality Division School, Bergen, Vestland
  - Haukeland University Hospital, Bergen